CLINICAL TRIAL: NCT04126993
Title: Anti-PD-1 Antibody SHR-1210 (Camrelizumab) Combined With Apatinib Mesylate in the Treatment of Unresectable Sarcoma With Chemotherapy Failure: an Open, Non-randomized Phase II Clinical Study
Brief Title: Study of SHR-1210 Combined With Apatinib in the Treatment of Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2019144
Record Dates: First submitted 2019-09-29; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-09

CONDITIONS: Sarcoma
Keywords: SHR-1210; Camrelizumab; Apatinib; Sarcoma; Jilong Yang
MeSH Terms: conditions — Sarcoma | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab+ Apatinib test group (Experimental): Camrelizumab intravenous injection once every three weeks, Apatinib 500 mg is administered orally daily, until disease progression or untolerable toxicity.
  Interventions: Drug: Camrelizumab,; Drug: Apatinib
- Apatinib single drug control group (Active Comparator): Apatinib 500 mg is administered orally daily, until disease progression or untolerable toxicity.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Camrelizumab, — Camrelizumab+ Apatinib test group: intravenous injection once every three weeks, Apatinib 500 mg is administered orally daily, until disease progression or untolerable toxicity.
  Arms: Camrelizumab+ Apatinib test group
Drug: Apatinib — Apatinib single drug control group: Apatinib 500 mg is administered orally daily, until disease progression or untolerable toxicity.

SUMMARY:
To observe the effectiveness of SHR-1210 (Camrelizumab) combined with apatinib in the treatment of unresectable sarcoma patients with chemotherapy failure. The main observations were progression-free survival (PFS) and progression-free control rate (PFR), followed by objective response rate (ORR) (CR+PR), disease control rate (DCR) (CR+PR+SD), and overall survival (OS).

To observe the safety of SHR-1210 (Camrelizumab) combined with apatinib in the treatment of sarcoma

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily join the study, sign informed consent, and have good compliance；
* Pathologically confirmed patients with unresectable sarcoma (except GIST), clinical stage using the American Cancer Research Joint Committee (AJCC) TNM staging criteria. At least 1 double-path measurable lesion according to CT or MR I;
* At least one chemotherapy regimen (containing an anthracycline) was used to treat patients with disease progression or intolerance according to the solid tumor efficacy evaluation criteria (RECIST 1.1);
* Clear cell sarcoma, alveolar soft tissue sarcoma can be directly into the group without chemotherapy;
* 14~75 years old, PS score: 0~2; expected survival period is more than 3 months;
* All acute toxic reactions caused by previous anti-tumor treatment or surgery are relieved to 0-1 before screening (according to NCI CTCAE version 4.03) or to the level specified by the enrollment/exclusion criteria (alopecia, etc. Except for toxicity that does not pose a safety risk to the subject);
* There are sufficient organ and bone marrow functions, defined as follows:

  * Blood routine (no blood transfusion within 14 days before treatment, no use of G-CSF, no use of drugs to correct), Neutrophil count (ANC) ≥ 1,500/mm3 (1.5 × 109/L); Platelet count (PLT) ≥ 100,000/mm3 (100 × 109/L); Hemoglobin (Hb) ≥ 9 g/dL (90 g/L);
  * Blood chemistry, Serum creatinine (Cr) ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance (Cockroft-Gault formula) ≥ 60 ml / min; Total bilirubin (TBIL) ≤ 1.5 × ULN; Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels ≤ 2.5 × ULN, liver metastases should be ≤ 5 × ULN;
  * Coagulation, International normalized ratio (INR) ≤ 1.5, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN;
  * Urine routine, Urine protein <2+; if urine protein ≥ 2+, 24-hour urine protein quantitation shows that the protein must be ≤ 1g;
  * Thyroid function, Thyroid stimulating hormone (TSH) ≤ ULN; if abnormalities should be considered T3 and T4 levels, T3 and T4 levels can be selected;
* Female subjects of childbearing age must undergo a serum pregnancy test within 7 days prior to treatment and the results are negative, and are willing to use a medically recognized effective contraceptive measure during the study period and within 3 months after the last administration of the study drug (eg: Intrauterine devices, contraceptives or condoms; for male subjects whose partners are women of childbearing age, surgical sterilization is required, or an effective method of contraception is recommended during the study period and within 3 months after the last study administration;
* With my consent and signed informed consent, I am willing and able to follow planned visits, research treatments, laboratory tests and other testing procedures.

Exclusion Criteria:

* The following treatments were received within 4 weeks of treatment:

  * Radiotherapy, surgery, chemotherapy, immunization or molecular targeted therapy for tumors; Other clinical research drugs; Vaccination live attenuated vaccine;
* Previously received treatment with PD-1/PD-L1/CTLA-4 antibody or VEGFR single target/multi-target inhibitor;
* Surgery and/or radiation therapy for soft tissue sarcomas is planned during the study (regardless of <5% of the bone marrow area);
* Imaging diagnosis of central nervous system tumors;
* Immune-suppressing drugs have been used within 14 days prior to initiation of treatment, excluding nasal and inhaled corticosteroids or physiological doses of systemic steroid hormones (That is, no more than 10 mg / day of prednisolone or equivalent physiological dose of other corticosteroids);
* There is any active autoimmune disease or a history of autoimmune disease (Including but not limited to: Autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism; Subjects with vitiligo or asthma that have been completely relieved in childhood and currently do not require medical intervention may be included, or a history of allogeneic organ transplantation or a history of allogeneic hematopoietic stem cell transplantation);
* Severe infections (such as intravenous infusion of antibiotics, antifungal or antiviral drugs) within 4 weeks prior to treatment, or unexplained fever >38.5 °C during screening/first administration;
* High blood pressure, and excellent control without antihypertensive medication (systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg)
* There are significant clinically significant bleeding symptoms or clear bleeding tendency within 3 months before treatment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ++ and above, vasculitis, etc. Or venous/venous thrombosis events occurring within 6 months prior to treatment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism; or require long-term anticoagulant therapy with warfarin or heparin, or long-term antiplatelet therapy (aspirin ≥ 300 mg / day or clopidogrel ≥ 75 mg / day);
* There were active heart disease in the 6 months before treatment, including myocardial infarction, severe/unstable angina. Echocardiography left ventricular ejection fraction <50%, poorly controlled arrhythmia (including QTcF interval men > 450 ms, women > 470 ms);
* Any other malignant tumor was diagnosed within 3 years prior to treatment, except for adequately treated basal cells or squamous cell skin cancer or cervical carcinoma in situ;
* It is known to be allergic to the study drug or any of its excipients; or to have a severe allergic reaction to other monoclonal antibodies;
* Human immunodeficiency virus (HIV) infection, active hepatitis B (HBV-positive and HBV DNA ≥ 500 IU/ml), Hepatitis C (positive hepatitis C antibody and higher detection limit of HCV-RNA than analytical methods);
* At the discretion of the investigator, there are concomitant diseases (such as poorly controlled hypertension, severe diabetes, neurological or psychiatric disorders, etc.) that seriously compromise the safety of the subject, may confuse the findings, or affect the subject's completion of the study. Any other situation.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Within 2 years
  PFS is defined as the length of time from random assignment to disease progression or to death resulting from any cause other than the progress.

SECONDARY OUTCOMES:
Disease control rate (DCR） | Within 2 years
  nvestigators will assess treatment response according to Response Evaluation Criteria in Solid Tumors 1.1（RECIST1.1）
Objective tumor response rate (ORR) | Within 2 years
  ORR is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response as best overall response according to radiological assessments.
Overall survival(OS) | Within 3 years
  OS is defined as the length of time from random assignment to death or to last contact.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Hospital & Institute, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol